CLINICAL TRIAL: NCT02478268
Title: Using MRI to Visualize Regional Therapy Response in Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bastiaan Driehuys (Other)
Collaborators: University of Wisconsin, Madison (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Bastiaan Driehuys, Associate Professor of Radiology, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00060259; R01HL126771 (NIH)
Record Dates: First submitted 2015-06-16; First posted 2015-06-23 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: idiopathic pulmonary fibrosis; xenon gas
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients with idiopathic pulmonary fibrosis (Active Comparator)
  Interventions: Drug: Hyperpolarized 129-Xenon gas; Device: MRI
- Healthy volunteers (Active Comparator)
  Interventions: Drug: Hyperpolarized 129-Xenon gas; Device: MRI

INTERVENTIONS:
Drug: Hyperpolarized 129-Xenon gas — Hyperpolarized xenon will be administered in multiple doses in volumes up to 25% of subject TLC followed by a breath hold of up to 15 seconds. Subsequent 129Xe doses will only be administered once the subject is ready to proceed.
  Other Names: Hyperpolarized 129Xe
Device: MRI — Conventional 1H MRI will be used to provide anatomical reference scans, as well as pulmonary perfusion.

SUMMARY:
The purpose of this study is to determine whether magnetic resonance imaging (MRI) using inhaled hyperpolarized 129Xe gas, and conventional contrast can help visualize impaired lung function and detect changes over time in patients receiving treatment as well as those who don't. 129Xe is a special type of xenon gas and when inhaled during MRI may be able to show areas of abnormal thickening of parts of the lungs. These images combined with images taken with injected contrast agents or other types of MRI may provide a better way to look at lung structure and function in patients with IPF. The ultimate goal is to predict how a particular patient might respond to a particular therapy and to observe such responses earlier than conventional tests. The investigators anticipate that the images acquired in this study will provide more specific information about lung disease than standard lung function tests. The use of 129Xe MRI is investigational. "Investigational" means that these tests have not yet been approved by the US Food and Drug Administration and are being tested in research studies like this one. In addition, standard MRI with contrast is not typically done as standard of care for monitoring progression of IPF, therefore, its use in this study is also considered investigational.

Healthy volunteers are being asked to participate in this study because the investigators need to develop a database of functional images that are representative of healthy lungs.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteer (technical optimization)
2. Outpatients of either gender, age > 18.
3. Willing and able to give informed consent and adhere to visit/protocol schedules. (Consent must be given before any study procedures are performed.)
4. Clinical diagnosis of IPF by established means

Exclusion Criteria:

1. Subject is less than 18 years old
2. MRI is contraindicated based on responses to MRI screening questionnaire
3. Subject is pregnant or lactating
4. Respiratory illness of a bacterial or viral etiology within 30 days of MRI
5. Subject has any form of known cardiac arrhythmia
6. Subject does not fit into 129Xe vest coil used for MRI
7. Subject cannot hold his/her breath for 15 seconds
8. Subject deemed unlikely to be able to comply with instructions during imaging
9. Recent exacerbation (within 30 days) defined by the need for antibiotics and/or systemic steroids
10. Medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-05; Primary Completion 2020-09-26 (Actual); Study Completion 2020-09-26 (Actual)

PRIMARY OUTCOMES:
Change in lung function as measured by ventilation defect percentage (VDP) | 12 months
  We expect that 129Xe ventilation defect percentage, and 129Xe ventilated lung volume measured 3 months after baseline, will predict CT progression observed 12 months from baseline

SECONDARY OUTCOMES:
Change in lung function as measured by gas exchange defect percentage (EDP) | 12 months
  Although the study is powered on ventilation defect percentage, we expect regional gas exchange defects to be a more sensitive marker of progression

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Mammarappallil, M.D., Principal Investigator — Duke University; Bastiaan Driehuys, Ph.D., Study Director — Duke University; Sean B Fain, Ph.D., Study Director — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - University of Wisconsin Madison, Madison, Wisconsin